CLINICAL TRIAL: NCT06939088
Title: Effect of Tirzepatide on Alcohol Intake and Reward Processing in Patients Diagnosed With Schizophrenia and Alcohol Use Disorder
Brief Title: Effects of Tirzepatide on Alcohol Intake in Patients Diagnosed With Schizophrenia and Alcohol Use Disorder
Acronym: DUALPSYCHIATRY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSc, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The DUALPSYCHIATRY study; U1111-1312-8134 (Registry Identifier: Universal Trial Number); 2024-518608-28-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse/Dependence; Alcohol Dependence; Alcoholism; Schizophrenia Disorders; Schizophrenia and Disorders With Psychotic Features; Schizophrenia and Schizophrenia Spectrum Psychosis; Schizophrenia
Keywords: GLP-1; Glucagon-like peptide 1; fMRI; GIP; Glucose-dependent Insulinotropic Polypeptide; Tirzepatide; Mounjaro(R); schizophrenia; alcohol; alcohol use disorder; dual diagnosis
MeSH Terms: conditions — Alcoholism; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Tirzepatide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide once-weekly s.c.titrated to a maximum dose of 15 mg
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Saline s.c. once-weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Once weekly injections s.c. with tirzepatide (Mounjaro(R))
  Other Names: Mounjaro
  Arms: Tirzepatide
Drug: Placebo — Once weekly injections s.c. with placebo (BD Posiflush)
  Other Names: BD Posiflush (saline)
  Arms: Placebo

SUMMARY:
Glucagon-like peptide-1 receptor agonists (GLP-1RAs), approved for the treatment of type 2 diabetes and obesity, have shown promise as a novel treatment for alcohol use disorder (AUD). This study aims to investigate whether the Glucose-dependent Insulinotropic Polypeptide/GLP-1RA tirzepatide will reduce alcohol consumption in patients with a dual diagnosis of AUD and schizophrenia, a population in dire need of improved treatment options. To further investigate the neurobiological underpinnings of a potential dampening effect on alcohol consumption, functional magnetic resonance imaging (fMRI) brain scans will be applied.

The key anticipated outcomes include:

* decreased alcohol consumption and
* reduced alcohol cue-induced brain activity in the GIP/GLP-1-treated patient group compared with the placebo group. To the best of the investigators knowledge, this has never been examined before.

DETAILED DESCRIPTION:
The study is a randomised (1:1), double-blinded, placebo-controlled clinical trial including 26 weeks of treatment investigating whether tirzepatide vs placebo can reduce the number of heavy drinking days in patients with comorbid diagnoses of schizophrenia and AUD. The primary endpoint will be evaluated after 16 weeks of treatment. The study will conclude after a post-intervention follow-up 14 weeks after last treatment at week 40 of the study.

108 participants will be included. Alcohol consumption and secondary endpoints will be assessed at weeks 0, 4, 8, 12, 16, 20, 26, and 40, and all patients will be offered 6 sessions of supportive therapy, while participating in the study.

The randomisation and administration of the weekly injections (tirzepatide/placebo) will be administered by an unblinded staff not involved in other trial activities. All patients will be blindfolded when receiving the injections. Eligible patients (n=50) will have an fMRI brain scan performed at baseline and in week 16. Blood tests for safety measures and secondary endpoint-measures will be performed at weeks 0, 16, 26, and 40.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: The patient must provide both oral and written informed consent.
* Diagnosis:

  * Diagnosed with alcohol dependence according to the International Classification of Diseases, 10th Edition (ICD-10), and alcohol use disorder as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
  * Diagnosed with schizophrenia spectrum disorder according to ICD-10 and DSM-5
* AUDIT Score: Alcohol Use Disorder Identification Test (AUDIT) score greater than 15.
* Body Mass Index (BMI): BMI of 23 kg/m² or higher.
* Age Range: Between 18 and 70 years old (inclusive).
* Heavy Alcohol Consumption: Defined as 4 or more heavy drinking days within a consecutive 21-day period during the 28 days preceding the baseline evaluation. The 21-day period will be selected based on the largest total alcohol consumption and the greatest number of heavy drinking days within the 28-day timeframe. This will be assessed using the Timeline Followback (TLFB) method. Heavy drinking days are defined as days with an alcohol intake of 4 or more units (48 g of alcohol) for women and 5 or more units (60 g of alcohol) for men.

Exclusion Criteria:

* Intellectual Disability: individuals with a diagnosis of intellectual disability.
* Acute Psychosis: Acute exacerbation of psychosis, as indicated by a score of 6 or 7 on the Clinical Global Impression-Severity (CGI-S) scale.
* Coercive Measures: Current use of coercive measures, which includes individuals sentenced to treatment ('dom til behandling').
* Suicidal Behaviour: Evidence of current severe suicidal behaviour, as assessed by the investigator during clinical evaluation.
* History of Severe Alcohol Withdrawal: History of delirium tremens or alcohol withdrawal seizures.
* Severe Withdrawal Symptoms: Clinical Institute Withdrawal Assessment of Alcohol Scale, revised (CIWA-Ar) score greater than 9 at baseline examination.
* Severe Neurological Conditions: Presence of severe neurological diseases, including severe traumatic brain injury.
* Diabetes: Type 1 or 2 diabetes
* Pregnant or Potentially Pregnant Women: WOCBP who are pregnant, breastfeeding, intend to become pregnant within the next 6 months (including 16 weeks of treatment plus two months after discontinuation of semaglutide), or are not using a highly effective contraceptive method throughout the study period. Highly effective methods include combined hormonal contraception (oral, intravaginal, transdermal), progestogen-only hormonal contraception (oral, injectable, implantable), intrauterine device (IUD), intrauterine system (IUS), bilateral tubal occlusion, vasectomised partner, or sexual abstinence. WOCBP with a measured serum human chorionic gonadotropin (hCG) level greater than 3 U/L at inclusion will also be excluded.
* Liver Function: Impaired hepatic function, defined as liver transaminases greater than three times the upper limit of normal.
* Renal Function: Impaired renal function, indicated by an estimated glomerular filtration rate (eGFR) below 50 mL/min and/or plasma creatinine above 150 μmol/L.
* Pancreatic Function: History of acute or chronic pancreatitis or amylase levels more than twice the upper limit of normal.
* Thyroid Conditions: Previous medullary thyroid carcinoma (MTC) or a family history of MTC and/or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).
* Cardiac Issues: Decompensated heart failure (NYHA class III or IV), unstable angina pectoris, or myocardial infarction within the past 12 months.
* Uncontrolled Hypertension: Systolic blood pressure above 180 mmHg or diastolic blood pressure above 110 mmHg.
* Alcohol Use Disorder Medication: Use of medications for alcohol use disorder (e.g., disulfiram, naltrexone, acamprosate, nalmefene) within the 28 days prior to inclusion as recorded in the Timeline Followback (TLFB) schedule.
* Investigational Drugs: Receipt of any investigational drug within the past three months.
* Weight-Lowering Medications: Use of other weight-lowering pharmacotherapy in the past three months.
* Allergic Reactions: Hypersensitivity to the active substance or any of the excipients.
* Language Barriers: Inability to speak and/or understand Danish.
* Other Conditions: Any other condition that, in the investigator's opinion, may interfere with participation in the trial.

For the subgroup of participants undergoing brain scans:

* MRI Contraindications: any contraindications for MRI (e.g., magnetic implants, pacemaker, claustrophobia).
* Benzodiazepine Use: Intermittent use of benzodiazepines within 12 days prior to the scanning session is not allowed. However, regular use of a stable dose of benzodiazepines is permitted.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heavy drinking days | From baseline to 16 weeks of treatment
  The primary endpoint will be a change in alcohol consumption, measured as a per cent change in heavy drinking days after 16 weeks of treatment with tirzepatide or placebo, adjusted for the value at baseline (percentage points). Heavy drinking days will be registered using the Timeline-Follow-Back (TLFB) method including the last 21 consecutive days with the largest total alcohol intake and the greatest number of heavy drinking days within the 28 days preceding the evaluation. A heavy drinking day is defined as more than 60/48 grams (men/women) of alcohol in one day.

SECONDARY OUTCOMES:
Heavy drinking days | From baseline to 26 weeks of treatment and 14 weeks post-intervention
  Change in heavy drinking days measured using the TLFB method.
Total alcohol consumption | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Change in total alcohol consumption measured using the TLFB method.
Days without alcohol consumption | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Change in number of days without alcohol measured using the TLFB method.
World Health Organization (WHO) Risk Levels of Alcohol Consumption | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Change in WHO alcohol risk level measured using the TLFB method.
Penn Alcohol Craving Scale (PACS) score | From baseline to 16 and 26 weeks of treatment
  Change in Penn Alcohol Craving Scale (PACS) score. Minimum score = 0, maximum score =30. A high score means a worse outcome.
Alcohol Use Disorder Identification Test (AUDIT) score | From baseline to 16 and 26 weeks of treatment
  Change in AUDIT score. Minimum score = 0, maximum score =40. A high score means a worse outcome.
Drug Use Disorders Identification Test (DUDIT) score | From baseline to 16 and 26 weeks of treatment
  Change in DUDIT score. Minimum score = 0, maximum score =44. A high score means a worse outcome.
Drug use frequency | From baseline to 16 and 26 weeks of treatment
  Change in drug use frequency measured using the drug use frequency section of the DUDIT-extended
Preferred substance of use | From baseline to 16 and 26 weeks of treatment
  Change in preferred substance of use
Biomarkers of cannabis exposure | From baseline to 16 and 26 weeks of treatment
  Changes in biomarkers of recent cannabis exposure (blood 11-hydroxy-delta 9-tetrahydrocannabinol (11-OH-THC) and 11-nor-9-carboxy-delta 9-tetrahydrocannabinol (THCCOOH) levels)
The Patient Health Questionnaire (PHQ-9) | From baseline to 16 and 26 weeks of treatment
  Changes in PHQ-9
Fagerströms Test for Nicotine Dependence score | From baseline to 16 and 26 weeks of treatment
  Changes in smoking habits using the Fagerströms Test for Nicotine Dependence score
Number of cigarettes smoked per day | From baseline to 16 and 26 weeks of treatment
  Changes in average number of cigarettes smoked per day
Cotinine levels | From baseline to 16 and 26 weeks of treatment
  Change in blood cotinine levels
Blood parameters | From baseline to 16 and 26 weeks of treatment
  Changes in blood parameters (GGT, ALAT, MCV)
Liver fibrosis (FIB-4 score) | From baseline to 26 weeks of treatment
  Changes in FIB-4 score
Blood phosphatidyl ethanol (PEth) levels | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Changes in PEth levels
Glycaemic control parameters | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Changes in HbA1c levels
Blood pressure | From baseline to 16 and 26 weeks of treatment
  Change in blood pressure
Body weight | From baseline to 16 and 26 weeks of treatment and 14 weeks post-intervention
  Change in body weight
Waist circumference | From baseline to 16 and 26 weeks of treatment
  Change in waist circumference
fMRI alcohol cue-reactivity | From baseline to 16 weeks of treatment
  Changes in fMRI BOLD signals in response to alcohol cues in brain regions related to reward in a subgroup (n=50) of participants
WHO-5 Subjective Well-Being Index | From baseline to 26 weeks of treatment
  Changes in quality of life measured using the World Health Organization-Five Well-Being Index (WHO-5)
Global Assessment of Psychosocial Disability (GAPD) | From baseline to 26 weeks of treatment
  Changes in GAPD score
Positive and Negative Syndrome Scale (PANSS-6) | From baseline to 26 weeks of treatment
  Changes in symptom severity of schizophrenia measured using PANSS-6
Clinical Global Impression Severity Scale (CGI-S) | From baseline to 26 weeks of treatment
  Changes in CGI-S score
Proteomics | From baseline to 16 and 26 weeks of treatment
  Change in proteomics
Qualitative experience | From baseline to 16 weeks of treatment
  For a subgroup of participants (n=20), qualitative interviews will be performed after 16 weeks of treatment to evaluate qualitative differences in trial participation experiences between the intervention and placebo groups, which will be assessed as a secondary outcome.

OTHER OUTCOMES:
Safety Outcome | From baseline to 16 and 26 weeks of treatment
  Suicidal ideation measured using the Columbia Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, MD, DMSc, Professor, Principal Investigator — Mental Healt h Service Centre Copenhagen , Frederiksberg Hospital, NP Lab
Locations (2):
- Denmark (2):
  - Department of Psychiatry, Aalborg University Hospital, Aalborg, Denmark
  - Psychiatric Center Copenhagen, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable relevant requests, e.g. for meta-analyses or independent validations. IPD will be shared anonymized or de-identified to protect participants' privacy and in accordance with relevant regulations (GDPR).
Supporting Information: Study Protocol, SAP